CLINICAL TRIAL: NCT04470323
Title: Functional Exhaustion of T Cells in COVID19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebatallah Hassan, dr, Assiut University
Other Study IDs: T cells
Record Dates: First submitted 2020-07-12; First posted 2020-07-14 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: T Cell Deficiency
MeSH Terms: conditions — Thymic aplasia | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples from patients and healthy volunteers were supplemented with anticoagulants (EDTA-K2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19 patients: Patients admitted to Assiut university Hospitals diagnosed as COVID19 positive patients by PCR.
  Interventions: Diagnostic Test: Flow cytometry
- healthy volunteer: as negative control for each sample
  Interventions: Diagnostic Test: Flow cytometry

INTERVENTIONS:
Diagnostic Test: Flow cytometry — Lymphocyte subsets in peripheral blood were assessed by staining 50 µl of blood sample with 5 µl of Fluoroisothiocyanate (FITC)-conjugated- PD-1, phycoerythrin (PE)-conjugated-CD8, peridinium-chlorophyll-protein (Per-CP)-conjugated-CD4, Peridinium-chlorophyll-protein (Per-CP)-conjugated anti-CD3 and allophycocyanin (APC) conjugated anti-CD28.

SUMMARY:
The primary end-point of our prospective, observational study is to count T cells in patients with laboratory-confirmed COVID-19 and healthy controls. In addition, the expression of T cell exhaustion marker was measured in COVID-19 cases.

DETAILED DESCRIPTION:
COVID-19 caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has posed great threat to human health. T cells play a critical role in antiviral immunity but their numbers and functional state in COVID-19 patients remain largely unclear. The immune response against viral infections depends on the activation of cytotoxic T cells that can clear infection by killing virus-infected cells, so boosting the numbers and function of T cells in COVID-19 patients is critical for successful recovery. However, the factors which might cause the reduction in count, and the activation status of T cells in COVID-19 patients, remain uninvestigated. Thus demonstration of T cell exhaustion during COVID-19 infection suggest that more urgent, early intervention may be required in patients with low T lymphocyte counts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Covid-19 test positive; hospitalized subjects; both sexes; given informed consent.

Exclusion Criteria:

* no exclusion criteriae

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Assiut university Hospitals diagnosed as COVID-19 positive patients by PCR.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
CD4+ (T-helper cells) in COVID 19 patients and healthy volunteers. | Baseline
  Detection of the percentage of CD4+ (T-helper cells) in COVID 19 patients and healthy volunteers.
CD8+ (T-cytotoxic cells) in COVID 19 patients and healthy volunteers. | Baseline
  Detection of the percentage of CD8+ (T-cytotoxic cells) in COVID 19 patients and healthy volunteers .
Detect PD-1 on CD8+ and CD4+ cells in COVID 19 patients and healthy volunteers . | Baseline
  Detection of the percentage of expression of PD-1 on CD8+ and CD4+ cells in COVID 19 patient and healthy volunteers.
Detect CD28+ and CD3+ cells in COVID 19 patients and healthy volunteers. | Baseline
  Detection of the frequency of CD28+ and CD3+ cells in COVID 19 patients and healthy volunteers .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diao B, Wang C, Tan Y, Chen X, Liu Y, Ning L, Chen L, Li M, Liu Y, Wang G, Yuan Z, Feng Z, Zhang Y, Wu Y, Chen Y. Reduction and Functional Exhaustion of T Cells in Patients With Coronavirus Disease 2019 (COVID-19). Front Immunol. 2020 May 1;11:827. doi: 10.3389/fimmu.2020.00827. eCollection 2020. PMID 32425950
- [Background] Li CK, Wu H, Yan H, Ma S, Wang L, Zhang M, Tang X, Temperton NJ, Weiss RA, Brenchley JM, Douek DC, Mongkolsapaya J, Tran BH, Lin CL, Screaton GR, Hou JL, McMichael AJ, Xu XN. T cell responses to whole SARS coronavirus in humans. J Immunol. 2008 Oct 15;181(8):5490-500. doi: 10.4049/jimmunol.181.8.5490. PMID 18832706
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570